CLINICAL TRIAL: NCT00047606
Title: Phase 4 Study to Compare Two Different IOP Lowering Medications for the Treatment of Open Angle Glaucoma or Ocular Hypertension in Caucasian and Japanese Subjects C-02-32.
Brief Title: Phase 4 Study Comparing IOP Lowering in OAG or OH in Caucasian or Japanese Subjects C-02-32
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-02-32; C-02-32
Record Dates: First submitted 2002-10-08; First posted 2002-10-11 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2008-08

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: open-angle; glaucoma; ocular; hypertension; POAG; Iris; Pigmentation; Japanese
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension

INTERVENTIONS:
Drug: IOP Lowering Medications

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of two different IOP lowering medications after six weeks of treatment in Caucasian and Japanese subjects.

ELIGIBILITY:
Adults of Caucasian and Japanese Ethnicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2002-08; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)